CLINICAL TRIAL: NCT01659983
Title: Comparison of Surgical Site Infection Between Delayed Primary Closure Versus Primary Closure in Complicated Appendicitis: A Multicenter Randomized Controlled Trial
Brief Title: Efficacy Study of Delayed Primary Closure to Reduce Rate of Wound Infection in Complicated Appendicitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Thammasat Hospital (Unknown); Chonburi hospital (Other Government); Vachira hospital (Unknown); Pathumtani Hospital (Unknown); Lampang Hospital (Other); Surin Hospital (Unknown)
Responsible Party: Principal Investigator, Boonying Siribumrungwong, Section for Clinical Epidemiology and Biostatistics, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 04-55-18 ว
Record Dates: First submitted 2012-06-25; First posted 2012-08-08 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Surgical Site Infection
Keywords: complicated appendicitis; wound closure; infection
MeSH Terms: conditions — Surgical Wound Infection; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary wound closure (Experimental): A wound will be sutured immediately after the operative procedure uisng non-absorbable monofilament suture or stapler at intervals of one centimeter apart and 0.5 cm back from a wound edge.
  Interventions: Procedure: Primary wound closure
- Delayed primary wound closure (Active Comparator): A wound will be left open with saline-soaked gauze packing after the operative procedure and will be sutured around day 3 to 7 after operation
  Interventions: Procedure: Primary wound closure

INTERVENTIONS:
Procedure: Primary wound closure — A wound will be sutured immediately after the operative procedure uisng non-absorbable monofilament suture or stapler at intervals of one centimeter apart and 0.5 cm back from a wound edge.

SUMMARY:
Research hypothesis:

Does delayed primary wound closure after appendectomy in adults with complicated appendicitis reduce postoperative superficial surgical site infection compare to primary wound closure.

Study design:

This study is a multicenter randomized controlled trial of delay versus primary wound closure in complicated appendicitis.

Setting:

Thammasat Hospital, Ramathibodi Hospital, Chonburi Hospital, Chonpratarn Hospital, Vachira Hospital, and Pathumthani Hospital

Participants:

Adult patients age 18 years or older and non-pregnant in women who have been diagnosed as gangrenous or ruptured appendicitis.

Outcome:

Superficial surgical site infection

Period of study:

August 2012 - August 2014

ELIGIBILITY:
Inclusion criteria

1. Adult patients age 18 years or older
2. Have been diagnosed as gangrenous or ruptured appendicitis base on clinical criteria with the following conditions

   a.Gangrenous appendicitis i.Erythematous or swelling of appendix and ii.Appearance of necrotic wall (dark, grayish color) b.Ruptured appendicitis i. Erythematous or swelling of appendix and ii.Appearance of hole in an appendix or iii.Rupture of appendix during a procedure c.Appearance of frank pus
3. Non-immunocompromised hosts which include

   1. AIDS
   2. History of end-stage renal disease (ESRD)
   3. History of autoimmune disease (SLE)
   4. Taking immunosuppressive agents (e.g, steroids, Cyclophosphamide, Tacrolimus, Mycophenolate mofetil)
   5. Cirrhosis with ascites
   6. Morbid obesity (BMI > 40 kg/m2)
4. Non-pregnant women
5. Willing to participate and provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Superficial surgical site infection (SSI) | within 1 month after operation
  Superficial SSI, which will be diagnosed using the Center for Disease Control (CDC) criteria as follows:
  * Infection within 30 days and
  * Involves only skin and subcutaneous tissue of the incision and
  * One of the following:
    * Purulent drainage,
    * organism isolated from culture of fluid or tissue
    * one of the following signs or symptoms:
    * pain or tenderness;
    * localized, swelling, redness, or
    * heat And the superficial incision is deliberately opened by surgeon

SECONDARY OUTCOMES:
postoperative pain | within 3 days after operation
  • Postoperative pain will be assessed using visual analog scale (VAS, ranged from 0-10) at day 1 and 3
Quality of life | 1 month after operation
  Quality of life will be assessed using the Thai EQ5D questionnaires before an operation, days 3 and 1 month after operation
Cost of treatment | 1 month after operation
  Both direct and indirect costs of treatment will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Boonying Siribumrungwong, MD, Principal Investigator — Ramathibodi Hospital; Ammarin Thakkinstian, PhD, Study Chair — Ramathibodi Hospital; Patarawan Woratanarat, Study Chair — Ramathibodi Hospital; Borwornsom Leerapan, Study Chair — Ramathibodi Hospital; Jittunut Hawanon, Study Chair — Thammasat Hospital
Locations (7):
- Thailand (7):
  - Vachira hospital, Dusit, Bangkok
  - Department of Surgery, Ramathibodi Hospital, Rachatevi, Bangkok
  - Chonburi hospital, Meaung, Changwat Chon Buri
  - Surin hospital, Meung, Changwat Surin
  - Pathumtani hospital, Meung, Pathumtani
  - Thammasat hospital, Rangsit City Municipality, Patumtani
  - Lampang hospital, Meung

REFERENCES:
- [Derived] Noorit P, Siribumrungwong B, Thakkinstian A. Clinical prediction score for superficial surgical site infection after appendectomy in adults with complicated appendicitis. World J Emerg Surg. 2018 Jun 18;13:23. doi: 10.1186/s13017-018-0186-1. eCollection 2018. PMID 29946346